CLINICAL TRIAL: NCT01395706
Title: Determination of the Sensitifity of ICG Fluorescence Technique for the Detection of Sentinel Lymph Nodes in Breast Cancer - a Monocenter Prospective Open-label Clinical Trial
Brief Title: ICG Fluorescence Technique for the Detection of Sentinel Lymph Nodes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pulsion Medical Systems SE (Industry)
Responsible Party: Gabriela Pühler, PULSION Medical Systems SE
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PULSION-001
Record Dates: First submitted 2011-07-14; First posted 2011-07-15 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-07

CONDITIONS: Malignant Neoplasm of Breast
Keywords: Malignant Neoplasm of Breast; Sentinel lymph node detection; ICG fluorescence technique; Population of male and female patients with mamma carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ICG flourescence technique (Experimental): This is an uncontrolled, non-randomised, open-label, monocenter clinical trial. A total of n=125 subjects will participate in this clinical trial. No clinical trial participant will be allowed to be included in this trial more than once.
  Interventions: Procedure: ICG Fluorescence technique

INTERVENTIONS:
Procedure: ICG Fluorescence technique — This is an uncontrolled, non-randomised, open-label, monocenter clinical trial.
  A total of n=125 subjects will participate in this clinical trial. No clinical trial participant will be allowed to be included in this trial more than once.
  10 mg (5mg/ml)per injection are applicated
  Other Names: Indocyanine Green (ICG)

SUMMARY:
Objectives of Clinical Trial

The main objective of this clinical trial is to show the efficacy of fluorescence lymphangiography with indocyanine green (ICG) for the detection of sentinel lymph nodes.

DETAILED DESCRIPTION:
Considering the high diagnostic accuracy and less vulnerable staging and therapy procedures, SLNB has rapidly become the state of the art diagnostic for axillary staging in early breast cancer.

Prior surgery, the so called sentinel lymph nodes are detected, harvested and histopathologically examined. The histopathologic status of the sentinel node thereby accurately reflects the status of the remaining axillary nodes. The sentinel lymph node biopsy allows minimizing risks and burdens for patients who very likely have no metastasis in the axillary lymph nodes sparing the ALND and reducing the risk of surgery and postoperative lymph oedema for instance. Contrarily to former procedure where an axillary lymph node dissection (ALND) was done each time, an ALND now only follows if the detected sentinel lymph node is metastatic.

Routinely sentinel lymph nodes are mapped using radiocolloid tracers such as technetium, sometimes combined with a blue dye.

However the infrastructure for a radioactive tracing is complex and not available easily: special techniques and equipment for the manufacturing of the radiocolloid as well as training in the use with radioisotopes are needed. For example, the application of radioactive markers needs a ready access to a nuclear medicine department, a pre-operative visit and an effective coordination between the involved disciplinesis. As these radioisotopes are formed by specialised, rare industry facilities availability is heavenly dependend and lack of radioisotopes with shortages in diagnostic procedures has already been reported. Furthermore radiocolloid mapping is associated with radioactive exposure of the concerned patients and health workers and imposes problems with surgical waste disposal.

Novel methods for detecting sentinel lymph nodes which waive the pre-operative injection of the radioactive marker are currently investigated. One of these new methods is the application of a fluorescence marker for SLN detection.

In this clinical trial a novel method for detecting the sentinel lymph node using indocyanine green, a fluorescent molecule shall by investigated.

ELIGIBILITY:
Inclusion Criteria:

* Early breast cancer: histopathologically confirmed diagnosis, maximum tumour stage T1 and T2, therefore diameter < 5 cm, unifocal tumour or multifocal tumour Grading G1-G3, invasive ductal and / or invasive lobar carcinoma ≤ 5 cm diameter
* Indicated sentinel lymph node biopsy as part of the patient's routine management for breast cancer
* Age: 18 - 80 years, inclusive
* Gender: male and female
* BMI: ≤ 30
* Non-smoker (for at least the previous 3 months)
* General operability
* Intact site-specific anatomy at the concerned breast and /or axilla for ensuring an adequate lymphangiography
* Performance of investigations with radioactive traced iodide at least 1 week before and 1 week after ICG application
* No clinically significant findings in the routine blood examinations
* Female subjects with childbearing potential must have a negative pregnancy test prior Tc application and must be either at least two years postmenopausal or using a highly effective mean of birth control (birth control that, alone or in combination, result in a low failure rate of less than 1 percent per year when used consistently and correctly):
* hormonal method of contraception,
* surgical sterility,
* double barrier methods,
* intrauterine contraceptive device,
* lifestyle with a personal choice of abstinence,
* bilateral vasectomy of sexual partner at least 3 months prior to enrolment in combination with barrier methods
* Willing and able to complete screening and study procedures, as described in the protocol
* Signed written informed consent to participate in this clinical trial

Exclusion Criteria:

* Breast cancer: stage T3 or T4 carcinoma, inflammatory or exulcerated mamma carcinoma
* Former operation in axilla
* Any previous radiotherapy at the concerned breast and / or axilla and / or chestwall
* Definite lymph node metastases (ultrasound and / or fine-needle aspiration) (definite nodal positive patients in fine-needle aspiration)
* Contraindication for technetium imaging
* History of allergy or hypersensitivity against the investigational medicinal products (its active substance or ingredients)
* History of intolerability to ICG-Pulsion during a previous injection, as this may lead to serious anaphylactic reactions
* History of allergic diseases / hypersensitivities, unless the investigator considers the allergic disease as clinically irrelevant for the purpose of this clinical trial
* Allergy to iodine or to shellfish
* Any other contraindication to one of the investigational medicinal products as described in their Summary of Product Characteristics
* Apparent hyperthyroidism, autonomous thyroid adenoma, unifocal, multifocal or disseminated autonomies of the thyroid gland
* Advanced renal impairment (creatinine > 1,5mg/dl)
* Complete lymphatic obstruction
* All clinically relevant internal medicinal diseases, cardiac or renal that could impair the outcome of the clinical trial or that in the investigator's mind are not compatible with participation for medical reasons
* Acute inflammatory or febrile illness
* Evidence of local inflammation at the site of surgery
* Concurrent medication or any medication during the 2 weeks preceeding the enrolment which reduce or increase the extinction of ICG (i.e. anticonvulsants, haloperidol)
* Current or recent history of illicit drug or alcohol abuse, or dependence as defined as the continued use of alcohol or drugs despite the development of social, legal, or health problems
* Psychiatric or cognitive impairment that, in the opinion of the investigator, would interfere with the subject's ability to comply with the study requirements (e.g. Alzheimer's disease)
* Pregnancy, breastfeeding
* Inability to understand the nature and the extent of the trial and the procedures required
* Missing signed written informed consent to participate in the clinical trial
* Participation in a drug trial during the whole clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-02 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Sensitivity using ICG | 5 to 11 days
  Intraindividual: number of tumour-involved fluorescent positive sentinel lymph nodes / total number tumour-involved Technetium positive sentinel lymph nodes

SECONDARY OUTCOMES:
Specificity using ICG | 5 to 11 days
  Specificity using ICG:
  number of patients with fluorescent positive sentinel lymph nodes that are not tumour - involved / number of patients with Tc positive SLN
  False negative rate:
  Number of patients where no sentinel lymph node is detected with Tc but with ICG / total number of patients with at least one Tc positive SLN
  Detection rate for the SLN using the ICG fluorescence imaging method:
  number of patients with at least one fluorescent sentinel lymph node per total number of patients treated with ICG Safety and tolerability of the IMP

CONTACTS AND LOCATIONS:
Overall Officials: Diethelm Wallwiener, Prof. Dr., Principal Investigator — University Hospital Tuebingen, University Department of Gynecology and Obstetrics
Locations (1):
- University Department of Gynecology and Obstetrics, Tübingen, Germany